CLINICAL TRIAL: NCT00248651
Title: Antidepressant Therapy for Functional Dyspepsia
Brief Title: Functional Dyspepsia Treatment Trial
Acronym: FDTT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Yuri A. Saito Loftus, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-05 (DK065713); U01DK065713 (NIH); NCT00275626 (obsolete NCT alias)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-06

CONDITIONS: Dyspepsia and Other Specified Disorders of Function of Stomach
Keywords: Bloating; Early Fullness; Nausea; Upper Abdominal Discomfort; dyspepsia; stomach pain; stomach discomfort
MeSH Terms: conditions — Dyspepsia; Nausea; Abdominal Pain | interventions — Amitriptyline; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amitriptyline (Active Comparator): Amitriptyline capsule (50 mg) plus a placebo escitalopram tablet will be taken at night half an hour before bedtime. To maximize patient tolerability, in the first 2 weeks the dose of amitriptyline will be 25 mg and then the dose will be increased to 50 mg, but the 25 mg and 50 mg capsules will be indistinguishable to maintain blinding.
  Interventions: Drug: Amitriptyline
- Escitalopram (Active Comparator): Escitalopram tablet (10 mg) plus a placebo amitriptyline capsule will be taken by mouth at night half an hour before bedtime for 12 weeks.
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Placebo escitalopram tablets and placebo amitriptyline capsules will be taken by mouth half an hour before bedtime for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amitriptyline — 25 mg capsule by mouth at bedtime for two weeks, then 50 mg capsule by mouth at bedtime for 10 weeks. The drug will be provided in blister packs.
  Other Names: Elavil
  Arms: Amitriptyline
Drug: Escitalopram — 10 mg tablets by mouth at bedtime for 12 weeks. The drug will be provided in blister packs.
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Placebo — Placebo escitalopram and placebo amitriptyline will be manufactured to ensure all tablets and capsules will be indistinguishable, and provided in blister packs.
  Arms: Placebo

SUMMARY:
Functional dyspepsia is a common gastrointestinal disorder. Symptoms can include stomach pain or discomfort, bloating, fullness after eating meals, and nausea. These symptoms often interfere with school and work, and weight loss may occur due to dietary restrictions.

The hypothesis of this study was that antidepressant therapy is more effective than placebo in relief of the symptoms of functional dyspepsia, adjusting for psychological and psychiatric co-morbidity. The study also examined if antidepressant therapy reduces disability and improves quality of life in functional dyspepsia.

DETAILED DESCRIPTION:
The aims of this study were to:

1. Determine whether antidepressant therapy is more efficacious than placebo in relief of the symptoms of functional dyspepsia, adjusting for psychological and psychiatric co-morbidity. The investigators also planned to determine if antidepressant therapy reduces disability, improves quality of life and influences clinical response over 6 months after ceasing medication.
2. Determine if gastric emptying (motor dysfunction) and the nutrient drink test (a test that assesses gastric hypersensitivity and/or gastric accommodation) is altered by antidepressant therapy with a tricyclic or selective serotonin re-uptake inhibitors (SSRI), and whether subgroups with altered physiology are associated with treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Normal esophagogastroduodenoscopy (EGD) (no esophagitis, Barrett's esophagus, cancer, erosions, or ulcer disease) within the past 5 years
* Diagnosis of functional dyspepsia
* Patients may have failed to adequately respond to antisecretory therapy in the past for functional dyspepsia to be suitable; a good response to antisecretory therapy, which remains first line therapy, suggests underlying gastroesophageal reflux disease (GERD).

Exclusion Criteria:

* Any documented history of endoscopic esophagitis, or predominant heartburn or acid regurgitation, or these symptoms two or more times per week in the prior year, to exclude GERD.
* Those who have had an adequate response to antisecretory therapy according to the physician interview, to exclude patients with disease easy to control with first line therapy or misdiagnosed GERD.
* Any documented peptic ulcer disease.
* Regular use of non-steroidal anti-inflammatory drugs (except long term low dose aspirin ≤ 325 mg / day)
* Subjects undergoing psychiatric treatment, having a current history of drug or alcohol abuse, or currently taking psychotropic medication for depression or psychosis, or eating disorders
* A history of abdominal surgery except appendectomy, cholecystectomy or hysterectomy, tubal ligations, bladder slings, and vasectomies
* Subjects with concurrent major physical illness (including cardiac or liver disease, diabetes, inflammatory bowel disease, glaucoma, urinary retention, active thyroid disease, vasculitis, lactose intolerance explaining symptoms)
* Subjects whose literacy skills are insufficient to complete self report questionnaires.
* Pregnancy, or refusal to apply adequate contraceptive measures during the trial
* Subjects currently on antidepressant therapy will be excluded.
* Patients who score 11 or greater on the 7 questions related to depression of the Hospital Anxiety Depression Scale will be excluded. These patients will be encouraged to get follow up for depression.
* All eligible patients over age 50 will have an EKG before randomization. Those found to have significant arrhythmias, conduction defects or a previous myocardial infarction on EKG will be excluded. Anyone with QT prolongation will be excluded.

The following concomitant medications will be prohibited during the trial:

* Systemically acting cholinergics and anticholinergics (atropine, didinium bromide, propantheline)
* Prokinetics (e.g., metoclopramide, tegaserod)
* Macrolide antibiotics (e.g., erythromycin, azithromycin)
* Aspirin (> 325 mg/day)
* Spasmolytics (e.g., dicyclomine)
* Antidepressants other than study medications
* Serotonin enhancing drugs: monamine oxidase inhibitors, anticonvulsants, dextromethorphan.

Participants will be instructed to avoid grapefruit/grapefruit juice during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2006-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Earnest P Bouras, M.D., Principal Investigator — Mayo Clinic; John K. DiBaise, M.D., Principal Investigator — Mayo Clinic; Colin P Howden, M.D., Principal Investigator — Northwestern University Chicago; Charlene M Prather, M.D., Principal Investigator — St. Louis University; Nicholas J Talley, M.D.,Ph.D., Study Chair — Mayo Clinic; Brian E. Lacy, M.D., Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center; G. R. Locke, III, M.D., Principal Investigator — Mayo Clinic; Bincy P Abraham, M.D., M.S., Principal Investigator — Baylor College of Medicine; Hashem El-Serag, M.D., Principal Investigator — Baylor College of Medicine; Paul Moayyedi, M.D., Principal Investigator — McMaster University Centre, Hamilton, Ontario
Locations (8):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Northwestern University Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Baylor College of Medicine, Houston, Texas
- McMaster University Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Herrick LM, Camilleri M, Schleck CD, Zinsmeister AR, Saito YA, Talley NJ. Effects of Amitriptyline and Escitalopram on Sleep and Mood in Patients With Functional Dyspepsia. Clin Gastroenterol Hepatol. 2018 Mar;16(3):401-406.e2. doi: 10.1016/j.cgh.2017.10.021. Epub 2017 Dec 1. PMID 29199141
- [Derived] Talley NJ, Locke GR, Saito YA, Almazar AE, Bouras EP, Howden CW, Lacy BE, DiBaise JK, Prather CM, Abraham BP, El-Serag HB, Moayyedi P, Herrick LM, Szarka LA, Camilleri M, Hamilton FA, Schleck CD, Tilkes KE, Zinsmeister AR. Effect of Amitriptyline and Escitalopram on Functional Dyspepsia: A Multicenter, Randomized Controlled Study. Gastroenterology. 2015 Aug;149(2):340-9.e2. doi: 10.1053/j.gastro.2015.04.020. Epub 2015 Apr 25. PMID 25921377
- [Derived] Herrick LM, Locke GR 3rd, Schleck CD, Zinsmeister AR, Treder V, Talley NJ. Dyspepsia in the community: value of a community-based mailed survey to identify potential participants for a randomized clinical trial. Scand J Gastroenterol. 2015 Aug;50(8):959-64. doi: 10.3109/00365521.2014.980317. Epub 2015 Mar 11. PMID 25761431
- [Derived] Talley NJ, Locke GR 3rd, Herrick LM, Silvernail VM, Prather CM, Lacy BE, DiBaise JK, Howden CW, Brenner DM, Bouras EP, El-Serag HB, Abraham BP, Moayyedi P, Zinsmeister AR. Functional Dyspepsia Treatment Trial (FDTT): a double-blind, randomized, placebo-controlled trial of antidepressants in functional dyspepsia, evaluating symptoms, psychopathology, pathophysiology and pharmacogenetics. Contemp Clin Trials. 2012 May;33(3):523-33. doi: 10.1016/j.cct.2012.02.002. Epub 2012 Feb 10. PMID 22343090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment was during October 27, 2006 to February 11, 2013.
Period: Overall Study
Arm/Group | Amitriptyline | Escitalopram | Placebo
Started | 97 | 98 | 97
Completed 12 Weeks of Treatment | 78 | 66 | 75
Completed | 69 | 58 | 65
Not Completed | 28 | 40 | 32
Not completed — Withdrawal by Subject | 28 | 40 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amitriptyline | Escitalopram | Placebo | Total
Number analyzed (Participants) | 97 | 98 | 97 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (15) | 45 (15) | 45 (16) | 44 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 72 | 73 | 219
  Male | 23 | 26 | 24 | 73
Region of Enrollment [Number; unit: participants]
  United States | 94 | 94 | 96 | 284
  Canada | 3 | 4 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Self-Report of Adequate Relief of Dyspepsia (Yes/No) For at Least 50% of Weeks 3 -12 of Treatment
Description: The first two weeks of treatment were excluded to allow for establishment of steady state drug levels.
Time Frame: 3 weeks through 12 weeks
Population: The intent-to-treat analysis included all randomized subjects.
Measure: Number; unit: percentage of participants
Arm/Group | Amitriptyline | Escitalopram | Placebo
Number analyzed (Participants) | 97 | 98 | 97
percentage of participants | 53 | 38 | 40
Statistical Analysis 1: Comparison: Amitriptyline vs Escitalopram vs Placebo; Overall treatment effect from logistic regression model incorporating balancing factors. A p-value of <0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.05, ANCOVA

2. Secondary Outcome: Gastric Emptying Half-Time (T1/2)
Description: The time for half of the ingested solids or liquids to leave the stomach.
Time Frame: 12 weeks
Population: The intent-to-treat analysis included all randomized subjects.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Amitriptyline | Escitalopram | Placebo
Number analyzed (Participants) | 97 | 98 | 97
minutes | 117 (43) | 108 (36) | 115 (40)

3. Secondary Outcome: Maximum Tolerated Volume by Nutrient Drink Test
Description: The nutrient drink test for meal-induced satiety had subjects drink 120 ml of ENSURE every four minutes. Satiety scores were measured on a scale graded 0-5 (1, no symptoms; 5, maximum satiety). When a score of 5 was reached, the maximum tolerated volume intake was measured. Abnormal satiety was defined as inability to consume > 800 ml of Ensure.
Time Frame: 12 weeks
Population: The intent-to-treat analysis included all randomized subjects.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Amitriptyline | Escitalopram | Placebo
Number analyzed (Participants) | 97 | 98 | 97
ml | 764 (319) | 823 (391) | 839 (442)

4. Secondary Outcome: Dyspepsia-Specific Quality of Life
Description: The Nepean Dyspepsia Index (NDI) assessed quality of life. NDI scores are summarized into overall quality of life and 5 subscales: Interference, Knowledge/Control, Eating/Drinking, Sleep Disturbance, Work/Study. The scale consists of 25 items, yielding 5 sub-scales. Range 0-100, higher numbers indicate a greater quality of life.
Time Frame: 12 Weeks
Population: The intent-to-treat analysis included all randomized subjects.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Amitriptyline | Escitalopram | Placebo
Number analyzed (Participants) | 97 | 98 | 97
units on a scale
  Overall Quality of Life | 80.6 [76.2 to 85.0] | 82.8 [78.4 to 87.1] | 73.5 [69.1 to 77.8]
  Interference Subscale | 83.2 [78.3 to 88.2] | 82.8 [78.4 to 87.1] | 76.2 [70.9 to 81.5]
  Knowledge/Control Subscale | 78.2 [73.2 to 83.2] | 76.2 [71.3 to 81.1] | 72.9 [68.2 to 77.6]
  Eat/Drink Subscale | 72.4 [66.7 to 78.0] | 70.6 [65.4 to 75.6] | 64.8 [59.6 to 70.1]
  Sleep Disturbance Subscale | 86.3 [81.6 to 91.0] | 80.8 [75.2 to 86.3] | 76.4 [70.9 to 81.8]
  Work/Study Subscale | 86.9 [82.6 to 91.1] | 87.2 [83.5 to 90.9] | 79.7 [74.5 to 84.9]
Statistical Analysis 1: Comparison: Amitriptyline vs Escitalopram vs Placebo; Comparison between antidepressant arms and placebo for overall quality of life. A p-value of <0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.02, ANCOVA
Statistical Analysis 2: Comparison: Amitriptyline vs Escitalopram vs Placebo; Comparison between antidepressant arms and placebo for Eat/Drink subscale. A p-value of <0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.06, ANCOVA
Statistical Analysis 3: Comparison: Amitriptyline vs Escitalopram vs Placebo; Comparison between antidepressant arms and placebo for Interference subscale. A p-value of <0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.06, ANCOVA
Statistical Analysis 4: Comparison: Amitriptyline vs Escitalopram vs Placebo; Comparison between antidepressant arms and placebo for Sleep Disturbance subscale. A p-value of <0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.01, ANCOVA
Statistical Analysis 5: Comparison: Amitriptyline vs Escitalopram vs Placebo; Comparison between antidepressant arms and placebo for Work/Study subscale. A p-value of <0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.04, ANCOVA

ADVERSE EVENTS:
Arm/Group | Amitriptyline | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/98 | 0/97
Other Adverse Events (participants affected / at risk) | 29/97 | 28/98 | 20/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amitriptyline (N=97) | Escitalopram (N=98) | Placebo (N=97)
Abdominal Pain (Gastrointestinal disorders) | 5 | 5 | 1
Black Stools (Gastrointestinal disorders) | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 1 | 1 | 1
C. Difficile Infection (Gastrointestinal disorders) | 1 | 0 | 0
Change in appetite (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 5 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0
Heartburn (Gastrointestinal disorders) | 1 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal fluid (Gastrointestinal disorders) | 0 | 0 | 2
Liver function abnormality (Hepatobiliary disorders) | 1 | 1 | 0
Nausea/Vomiting (Gastrointestinal disorders) | 6 | 9 | 3
Anxiety (Nervous system disorders) | 2 | 6 | 4
Depression (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 11 | 1
Dream abnormalities (Nervous system disorders) | 1 | 0 | 0
Drowsiness or Somnolence (Nervous system disorders) | 14 | 10 | 5
Headache (Nervous system disorders) | 2 | 8 | 3
Insomnia (Nervous system disorders) | 2 | 5 | 1
Tingling (Nervous system disorders) | 1 | 1 | 1
Chest pain (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Vasovagal syncope (Cardiac disorders) | 0 | 1 | 1
Abrasion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 5
Decreased libido (Endocrine disorders) | 0 | 3 | 0
Enlarged thyroid (Endocrine disorders) | 0 | 1 | 0
Hot/cold sensitivity (Endocrine disorders) | 0 | 1 | 1
Ovarian cysts (Endocrine disorders) | 2 | 0 | 0
Bruising (Blood and lymphatic system disorders) | 0 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Edema (Metabolism and nutrition disorders) | 0 | 0 | 2
Weight gain (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0
Pain (other than back and pelvic) (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Pelvic pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Infectious (Ear and labyrinth disorders) | 1 | 0 | 0
Non-infectious (Ear and labyrinth disorders) | 2 | 2 | 1
Infectious (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1
Non-infectious (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Infection (Eye disorders) | 0 | 1 | 0
Non-infection (Eye disorders) | 1 | 0 | 0
Vision changes (Eye disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Prostate infection (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No